CLINICAL TRIAL: NCT05727969
Title: Effect Of Dexmedetomidine Infusion On Surgical Pleth Index In Pediatrics Undergoing Hypospadias Repair; A Prospective Observational Study
Brief Title: Dexmedetomidine Infusion and Surgical Pleth Index In Pediatrics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Hamed, Associate professor of anesthesia, Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: M637
Record Dates: First submitted 2023-01-24; First posted 2023-02-14 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Pain; Hypospadias
Keywords: Dexmedetomidine; Hypospadias; Postoperative analgesia; Surgical pleth index
MeSH Terms: conditions — Pain; Hypospadias | interventions — Dexmedetomidine; Ringer's Lactate; Solutions

STUDY DESIGN:
Intervention Model Description: The randomization will be computer generated random number and the randomization sequence will be kept hidden in sealed opaque envelopes just opened after recruitment and admittance to the operating room.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The group's allocations will be only blinded to assessors, data collectors, and parents of children
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Placebo Comparator): The control group, lactated ringer solution will be infused.
  Interventions: Drug: Lactated Ringer; Procedure: Hypospadias; Device: Surgical pleth index
- Dexmedetomidine group (Experimental): In the dexmedetomidine group, dexmedetomidine will be infused.
  Interventions: Drug: Dexmedetomidine; Procedure: Hypospadias; Device: Surgical pleth index

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine at a a rate of 0.5 μg/kg/hour will be infused with induction of anesthesia.
  Other Names: Precedex
  Arms: Dexmedetomidine group
Drug: Lactated Ringer — Lactated ringer solution at a a rate of 0.5 μg/kg/hour will be infused with induction of anesthesia.
  Other Names: Solution
  Arms: Control group
Procedure: Hypospadias — Children who will undergone hypospadias surgery
  Other Names: pediatric manuvere
Device: Surgical pleth index — The SPI value will be measured using Datex-Ohmeda (GE Healthcare,Madison,WI 53707-7550 USA) monitoring system.
  Other Names: SPI

SUMMARY:
This non-invasive dimensionless score index -SPI-reflects the Patients' sympathetic response to surgical stimulation. Its effectiveness in detecting the balance between nociceptor activation and analgesia was not only reported but also, was reported to be superior to the other parameters like blood pressure and heart rate. SPI value is correlated to pain and ranges from 0 to 100, higher values indicate strong surgical stimulus. Its value is obtained from photoplethysmographic amplitude (PPGA) and heart rate (HR) data from pulse oximetry measurement.

Prediction of the severity of postoperative pain using SPI in both adults and children has been reported by several studies. So, the authors hypothesize that dexmedetomidine infusion without giving a bolus dose may affect the SPI in pediatrics undergoing hypospadias repair.

DETAILED DESCRIPTION:
After obtaining Fayoum University's ethical committee permission and as well as the informed consent from the parents, 90 patients aged 1 to 7 years old scheduled for hypospadias repair will be randomly assigned into 2 groups.

Preoperative Assessment:

All patients will be assessed clinically and investigated for exclusion of any of the above-mentioned contraindications.

Perioperative Management:

Patients will receive no premedication. After entering the Operating room, All patients will be monitored using surgical pleth index, arterial blood pressure, pulse oximetry, and electrocardiography. The SPI value will be measured using Datex-Ohmeda (GE Healthcare,Madison,WI 53707-7550 USA) monitoring system.

Inhalational induction of general anesthesia (GA) will be performed with a face mask using sevoflurane 8% and 50% oxygen in the air, and then an intravenous (IV) cannula will be inserted.

Fentanyl will be administered intravenously at 1 μg/kg, atracurium 0.5 mg/kg and an endotracheal tube will be used to secure the airway.

Anesthesia will be maintained with 1% isoflurane, 50% oxygen in the air, and atracurium infusion (0.10 mg/kg).

During the operation, bradycardia is defined as a 30% decrease from the baseline HR, and hypotension is defined as a 30% decrease from the baseline MAP. In these cases, 0.01 mg/kg of atropine and 0.1 mg/kg of ephedrine, respectively, will be given intravenously. Additionally, tachycardia is defined as a 30% increase from the baseline HR, and hypertension is defined as a 30% increase from the baseline MAP. If either of these occurred, 0.1 μg/kg of fentanyl was given intravenously, and then the incidence was calculated and analyzed.

At the end of the surgery, acetaminophen 15 mg/kg IV will be administered to all patients. After completion of the surgical procedure and emergence from anesthesia, the patient will be referred to PACU. Quality of analgesia will be assessed using a face, legs, activity, cry, consolability (FLACC scale) at PACU discharge and 2, 4, 6, 12, and 24 hours postoperatively. Diclofenac sodium 1 mg/kg rectally will be given as rescue analgesia for patients in all study groups in PACU if the FLACC scale > 4. Nurses will be informed about the pain evaluation, to give the patients oral paracetamol 30 mg/kg. The data collectors from nurses will record data. The depth of sedation will be assessed using Ramsy sedation score (RSS) at PACU discharge and 2 hours postoperative by the investigators.

The patient will be discharged from PACU using The Modified Aldrete Score system after an assessment of the patient's activity, respiration, blood pressure, consciousness, and color, A score ≥ 9 is required for discharge from the PACU.

Adverse events like bradycardia hypotension excessive sedation respiratory depression postoperative agitation nausea and vomiting will be recorded during the first 24 hours.

Statistical analysis

* Sample size calculation was done using IBM SPSS version 29 for Windows. A total of 45 children per group are needed to be able to detect an expected difference in the SPI based on previous research.This sample size was estimated using a power of 80% and alpha of 0.05.
* Descriptive statistics for the variables will be presented in the form of mean with standard deviation or median with interquartile range for numeric variables, while frequencies and percentages will be used for categorical variables. Comparison of the two groups will be done after testing for normality of the distribution using Shapiro-wilk test. The analysis will be done using the independent samples t test or using the non-parametric Mann Whitney test for numerical variables. Categorical variables will be compared using Chi Square test or Fisher's exact test. IBM SPSS version 28 for Windows software will be used for the analysis. A p-value of < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Age 1-7years.
* ASA physical status I-II.
* Hypospadias surgery.

Exclusion Criteria:

* Children having a history of mental retardation.
* Developmental delay.
* Allergic to dexmedetomedine.
* Neuraxial anesthesia.
* Cardiovascular disease.

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Surgical pleth index number | 1 minute at end of the operation after skin closure.
  from 0 to 100, higher values indicate strong surgical stimulus

SECONDARY OUTCOMES:
Surgical pleth index number | 1 minute before induction of anesthesia.
  from 0 to 100, higher values indicate strong surgical stimulus
Surgical pleth index number | 1 minute after insertion of endotracheal tube.
  from 0 to 100, higher values indicate strong surgical stimulus
Surgical pleth index number | 1 minute after beginning of surgery with skin incision.
  from 0 to 100, higher values indicate strong surgical stimulus
Surgical pleth index number | 5 minutes after recovery at post anesthesia care unit.
  from 0 to 100, higher values indicate strong surgical stimulus
Mean arterial blood pressure | 5 minutes after recovery at post anesthesia care unit.
  in mmHg
Mean arterial blood pressure | 1 minute before induction of anesthesia.
  in mmHg
Mean arterial blood pressure | 1 minute after beginning of surgery with skin incision.
  in mmHg
Heart rate | 1 minute after beginning of surgery with skin incision.
  beat/minute
Heart rate | 1 minute before induction of anesthesia.
  beat/minute
Heart rate | 5 minutes after recovery at post anesthesia care unit.
  beat/minute
Heart rate | 1 minute at end of the operation after skin closure.
  beat/minute
Mean arterial blood pressure | 1 minute at end of the operation after skin closure.
  mmHg
Need of vasoactive drugs | 1minute after infusion until end of surgery
  Yes or no
FLACC pain score | 5 minutes after recovery in postanesthesia care unit
  F:face - L:legs - A:activity - C:cry - C:consolability for description of pain degree in children
FLACC pain score | 2 hours after recovery in postanesthesia care unit
  F:face - L:legs - A:activity - C:cry - C:consolability for description of pain degree in children
Ramsay sedation score | 5 minutes after recovery in postanesthesia care unit
  0:5 with 0:deeply sedation to 5:no sedation
Ramsay sedation score | 2 hours after recovery in postanesthesia care unit
  0:5 with 0:deeply sedation to 5:no sedation
FLACC pain score | 4 hours after discharge from recovery
  F:face - L:legs - A:activity - C:cry - C:consolability for description of pain degree in children
FLACC pain score | 6 hours after discharge from recovery
  F:face - L:legs - A:activity - C:cry - C:consolability for description of pain degree in children
FLACC pain score | 12 hours after discharge from recovery
  F:face - L:legs - A:activity - C:cry - C:consolability for description of pain degree in children
FLACC pain score | 24 hours after discharge from recovery
  F:face - L:legs - A:activity - C:cry - C:consolability for description of pain degree in children
Surgical time | 1 minute after skin
  from when the surgeon of record starts the procedure until complete skin closure in minutes
Anesthesia time | 5 minutes after insertion of endotracheal tube
  from the start of anesthesia to the end of an anesthesia service in minutes
Total opioid consumption | 24 hours after operation
  in milligram
Time of 1st analgesia dose | 24 hours postoperatively
  time when first analgesic drug is injected for pain (in hours)
Total non-steroidal consumption | 24 hours postoperatively
  time when first usage of non-steroidal anti-inflammatory drug is injected for pain (in hours)
Extubation time | 2 minutes after removal of endotracheal tube
  time from the end of surgery to airway extubation (in minutes)

OTHER OUTCOMES:
Age | 1 hour preoperatively
  in years
American society of anesthesiology classification | 1 hour preoperatively
  Either I: normal healthy or II: mild systemic disease

CONTACTS AND LOCATIONS:
Overall Officials: Safaa G Megahed, MD, Study Director — Fayoum University; Omar S Mahmoud, MD, Study Director — Fayoum University
Locations (1):
- Fayoum University hospital, El Fayoum Qesm, Faiyum Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huiku M, Uutela K, van Gils M, Korhonen I, Kymalainen M, Merilainen P, Paloheimo M, Rantanen M, Takala P, Viertio-Oja H, Yli-Hankala A. Assessment of surgical stress during general anaesthesia. Br J Anaesth. 2007 Apr;98(4):447-55. doi: 10.1093/bja/aem004. Epub 2007 Feb 28. PMID 17329347
- [Background] Hamunen K, Kontinen V, Hakala E, Talke P, Paloheimo M, Kalso E. Effect of pain on autonomic nervous system indices derived from photoplethysmography in healthy volunteers. Br J Anaesth. 2012 May;108(5):838-44. doi: 10.1093/bja/aes001. Epub 2012 Feb 26. PMID 22369767
- [Background] Constant I, Sabourdin N. Monitoring depth of anesthesia: from consciousness to nociception. A window on subcortical brain activity. Paediatr Anaesth. 2015 Jan;25(1):73-82. doi: 10.1111/pan.12586. Epub 2014 Nov 20. PMID 25410376